CLINICAL TRIAL: NCT06784375
Title: Personalized Nutrition Using Continuous Glucose Monitoring to Improve Outcomes in Type 2 Diabetes Mellitus
Brief Title: Personalized Nutrition for Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MED-2024-31907
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Nutrition; CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Unblinded CGM/Nutrition Therapy (Experimental)
  Interventions: Behavioral: Unblinded CGM/Nutrition Therapy
- Blinded CGM/Nutrition Therapy (Experimental)
  Interventions: Behavioral: Blinded CGM/Nutrition Therapy
- Unblinded CGM/No Nutrition Therapy (Experimental)
  Interventions: Behavioral: Unblinded CGM/No Nutrition Therapy
- Blinded CGM/No Nutrition Therapy (Experimental)
  Interventions: Behavioral: Blinded CGM/No Nutrition Therapy

INTERVENTIONS:
Behavioral: Unblinded CGM/Nutrition Therapy — Personalized nutrition counseling based on CGM data
  Arms: Unblinded CGM/Nutrition Therapy
Behavioral: Blinded CGM/Nutrition Therapy — Standard nutrition education which does not incorporate CGM data
  Arms: Blinded CGM/Nutrition Therapy
Behavioral: Unblinded CGM/No Nutrition Therapy — CGM and general diabetes education (no nutrition education)
  Arms: Unblinded CGM/No Nutrition Therapy
Behavioral: Blinded CGM/No Nutrition Therapy — General diabetes education (no nutrition education)
  Arms: Blinded CGM/No Nutrition Therapy

SUMMARY:
This project will compare medical nutrition therapy personalized by continuous glucose monitor (CGM) feedback to control interventions in participants with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* previous diagnosis of T2DM
* HbA1c of 6.8-8.5%

Exclusion Criteria:

* type 1 diabetes mellitus
* treatment with insulin, sulfonylurea, or meglitinide
* use of nondiabetic medications that affect blood glucose control (such as corticosteroids)
* BMI <25 kg/m2 or <23 kg/m2 for participants who self-identify as Asian
* weight change >5 pounds in the 3 months prior to study enrollment
* estimated glomerular filtration rate <60 ml/minute/1.73 m2
* pregnancy or immediate plans to become pregnant 8) breastfeeding 9) anemia (which would affect measurement of HbA1c) 10) changes to glucose lowering medications, including change in dose, in the 3 months prior to enrollment 11) presence of any disease that would make adherence to the protocol difficult."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 12 weeks
  Measure of blood glucose control

CONTACTS AND LOCATIONS:
Overall Officials: Anne Bantle, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States